CLINICAL TRIAL: NCT04096768
Title: Combining Dexmedetomidine and Ketamine in Intensive Care Sedation: Efficacy and Safety
Brief Title: The Use of Ketamine and Dexmedetomidine in Intensive Care Sedation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lebanese American University Medical Center (Other)
Responsible Party: Principal Investigator, Fayez Abillama, MD, Intensive Care Medicine Physician, Lebanese American University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FA2.2016.R2.21/Jun/2019
Record Dates: First submitted 2019-09-15; First posted 2019-09-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: ICU Patients; Sedation
MeSH Terms: interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine + Ketamine (Experimental)
  Interventions: Drug: Dexmedetomidine; Drug: Ketamine
- Dexmedetomidine + Placebo (Placebo Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Comparing Dexmedetomidine + Ketamine versus Dexmedetomidine + Placebo for sedation in ICU patients
Drug: Ketamine — Comparing Dexmedetomidine + Ketamine versus Dexmedetomidine + Placebo for sedation in ICU patients
  Arms: Dexmedetomidine + Ketamine

SUMMARY:
The aim of the study is to compare the use of dexmedetomidine + ketamine with dexmedetomidine + placebo for sedation in ICU patients in terms of safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years old
* Admitted to Intensive care unit at LAUMCRH
* Need for sedation for at least 24 hours
* Informed Consent Form signed by patient or surrogate

Exclusion Criteria:

* Pregnant patients
* At risk of increased intracranial pressure
* Aortic dissection
* Acute coronary syndrome
* Hypertension (SBP > 180 mmHg)
* Chronic alcoholism
* Acute alcohol intoxication
* Alcohol withdrawal
* Refractory status epilepticus
* History of psychiatric disorder
* Known allergy or contraindication to use of dexmedetomidine or ketamine
* Baseline hypotension (MAP<65 mmHg)
* Baseline bradycardia (HR<48 bpm)
* Patients receiving neuromuscular blocking agents
* Patients requiring deep sedation as determined by the ICU attending

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-09-16 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Measuring blood pressure to assess hypotension when using a combination of the two drugs for sedation versus Dexmedetomidine and placebo only | Within 24 hours of drugs administration
  Measuring blood pressure to assess hypotension when using a combination of the two drugs for sedation versus Dexmedetomidine and placebo only

SECONDARY OUTCOMES:
Measuring the doses of dexmedetomidine and ketamine when combined and the doses of dexmedetomidine when used alone to achieve desired level of sedation | Within 24 hours of drugs administration
  Measuring the doses of dexmedetomidine and ketamine when combined and the dose of dexmedetomidine when used alone to achieve desired level of sedation

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese American University Medical Center- Rizk Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided